CLINICAL TRIAL: NCT06712186
Title: Title: the Effects of Dexmedetomidine on Hemodynamic Responses to Endotracheal Intubation in Hypertensive Patients Undergoing Surgery
Brief Title: Effect of Dexmedetomidine on Hemodynamic Response to Endotracheal Intubation in Hypertensive Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Warisha Ismail, Warisha Ismail Dr, FCPS I, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: App #0877-2023-LNH-ERC
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Elective Surgical Patient; Hypertensive Patients; Blood Pressure; Hypertensive Elderly Patients; Anxiolytic
Keywords: Laryngoscopy; Dexmedetomidine; Hemodynamic Response; Endotracheal intubation; Pressor response; Hypertension; Intubation; General anesthesia; a 2 agonist; Sedative; Anxiolytic
MeSH Terms: conditions — Hypertension | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group/Group D (Experimental): Intervention group: Group D patients will be administer 0.5 mcg/kg dexmedetomidine intravenously over 10 min preoperatively.
  Interventions: Drug: Dexmedetomidine Group / Group D
- Control group/Group C (Placebo Comparator): Control group: Group C patients will be administer the same volume of normal saline (also intravenously for 10 min)
  Interventions: Other: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Dexmedetomidine Group / Group D — In this study, the intervention involve administrating 0.5 mcg/kg of Inj dexmedetomidine intravenously over 10 min to patients in intervention group/group D 2 minutes prior to Endotracheal intubation using laryngoscopy aiming to asses its efficacy in attenuating the pressor response to laryngoscopy.
  Other Names: Dexemeditomidine
  Arms: Intervention group/Group D
Other: Normal Saline (Placebo) — The Placebo group / group C will be administer Normal Saline without any active medication over 10 min to patients, 2 minutes prior to Endotracheal intubation using laryngoscopy to compare its effect to those of Dexmedetomidine in attenuating the pressor response to laryngoscopy.
  Other Names: normal saline
  Arms: Control group/Group C

SUMMARY:
Dexmedetomidine, an alpha-2 adrenergic agonist, has been shown to provide several benefits during endotracheal intubation:

1. _Reduced anxiety and stress_: Dexmedetomidine's anxiolytic and sedative effects help reduce anxiety and stress associated with endotracheal intubation.
2. _Improved intubating conditions_: Dexmedetomidine can improve intubating conditions by reducing the incidence of coughing, bucking, and laryngospasm.
3. _Decreased hemodynamic responses_: Dexmedetomidine can attenuate the hemodynamic responses to intubation, including tachycardia, hypertension, and increased cardiac output.
4. _Increased ease of intubation_: Dexmedetomidine can facilitate smoother and easier intubation by reducing the need for additional anesthetics or muscle relaxants.

The physiological responses to dexmedetomidine during intubation include:

1. _Decreased heart rate_: Dexmedetomidine can cause a decrease in heart rate due to its effects on the sympathetic nervous system.
2. _Decreased blood pressure_: Dexmedetomidine can also cause a decrease in blood pressure due to its vasodilatory effects.
3. _Increased sedation_: Dexmedetomidine's sedative effects can help reduce anxiety and stress during intubation.
4. _Reduced respiratory rate_: Dexmedetomidine can cause a decrease in respiratory rate due to its effects on the respiratory centers in the brain.

The clinical benefits of dexmedetomidine during intubation include:

1. _Improved patient comfort_: Dexmedetomidine's sedative and anxiolytic effects can improve patient comfort during intubation.
2. _Reduced need for additional anesthetics_: Dexmedetomidine can reduce the need for additional anesthetics or muscle relaxants during intubation.
3. _Decreased risk of complications_: Dexmedetomidine's effects on hemodynamic responses and respiratory rate can decrease the risk of complications during intubation.

DETAILED DESCRIPTION:
General anesthesia during surgery produces a state of controlled unconsciousness during which the patient is unaware and insensitive to pain. Laryngoscopy and endotracheal intubation are mostly used to maintain airway while the patient is unconscious. Following the induction of anaesthesia, direct laryngoscopy and tracheal intubation are attributed to hemodynamic alterations brought on by sympathetic adrenergic outflow caused by laryngeal tissue stimulation, which may cause hypertension, tachycardia, arrhythmia, raised intracranial pressure, and intraocular pressure. The hemodynamic changes brought about by laryngoscopy and intubation were first described by Reid and Brace.This may be inconsequential in normal people but may lead to serious morbidity in patients with coexisting cerebrovascular or cardiovascular conditions.Patients undergoing treatment for hypertension have more pronounced hemodynamic responses to sympathetic stimulation.

Dexmedetomidine is a highly selective α-2 adrenoceptor agonist with a distribution half-life of approximately 6 minutes frequently used in anesthesia practice. With only minimal respiratory depression and cardiovascular stability, dexmedetomidine produces sedation, hypnosis, analgesia, anxiolysis, and sympatholysis. The central effects are due to the activation of α-2A receptors in locus coeruleus, and cardiovascular effects are due to a dose-dependent decrease in the central sympathetic outflow. The transient hypertensive response is seen initially due to its effects on α-2B receptors present in the vascular smooth muscle until there is a decrease in the central sympathetic outflow.

The study's main aim is to assess the effectiveness of using dexmedetomidine as a preventative measure to lessen the sympathetic response caused by tracheal intubation in hypertensive individuals.

The objective of the study is to compare mean attenuation of stress response between groups given dexmedetomidine versus Normal Saline among hypertensive patients undergoing general anaesthesia with endotracheal intubation. We want to compare the effect of Dexmedetomidine on MAP at 5 minutes after laryngoscopy.

The study design is Prospective double blind Randomized Controlled Trial and will be conducted in Department of Anesthesia, Liaquat National hospital.

The 60 patients from Anesthesia Preoperative Clinic will be randomly allocated to 2 groups by using a closed-envelope method-a control group (group C) that will receive normal saline and a comparative group (group D) that will receive dexmedetomidine. Group D patients (n = 30) will be administer 0.5 mcg/kg dexmedetomidine (PrecedexTM; Hospira Inc., Lake Forest, IL, USA) intravenously over 10 min. Group C patients will be administer the same volume of normal saline (also intravenously for 10 min). Saline and dexmedetomidine will be administer using a syringe pump by an anesthesiologist unaware of the study protocol. After completing the saline or dexmedetomidine administration, Propofol (1.5-2.5mg/kg) titrated to effect and Atracurium (0.5 mg/kg) will be administer. Two minutes after these administrations, endotracheal intubation will be perform using a laryngoscope. All intubations will be performed within <30 sec by one anesthesiologist. Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), and heart rate (HR) will be recorded in the ward just before departure to the operating room (baseline value), immediately after study drug administration, and at 1, 3, and 5 min after endotracheal intubation.The primary outcome is MAP at 5 min while HR, Systolic blood pressure and diastolic blood pressure are secondary outcome.

Data will be analyzed by using IBM SPSS Statistics version 26. Normality will be checked by Shapiro w\Wilk test.Stratification will be done with regards to age, weight and duration of hypertension, gender, comorbid other than hypertension and drug used as per need and post stratification independent t test/ Mann-Whitney U-test will be applied. P<0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA Grade II
* Age > 60 years
* Elective surgical procedures under GA.
* All patients with a diagnosis of hypertension for 6 months or more and undergoing treatment with antihypertensive medications.

Exclusion Criteria:

* Patient refusal
* ASA Grade III and IV
* Severely Hypovolemic state
* Emergency surgeries
* Body weight more than 20% of ideal body weight.
* Patients with known or unanticipated difficult intubation and those requiring more than 15 sec or two attempts at laryngoscopy
* Allergic to dexmedetomidine
* Non complaint hypertensive patients
* Patients with uncontrolled hypertension.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-22 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean Arterial Pressure (MAP) | At 5 minutes after laryngoscopy and endotracheal intubation.
  The primary outcome is to measure the change in Mean Arterial Pressure before endotracheal intubation and 5 minutes after intubation.
  An increase or decrease in MAP of 20 mmHg of patient's baseline MAP within 5 minutes of endotracheal intubation will be considered significant in our study.
  The focus is on whether Dexmedetomidine maintain MAP with 20mmhg of patient's baseline reading.

SECONDARY OUTCOMES:
Heart Rate (HR) | Baseline & 5 minutes
  A increase or decrease in HR of 20 bpm of patient's baseline HR within 5 minutes of endotracheal intubation will be considered significant in our study.
Blood pressure (BP) | Baseline & 5 minutes
  An increase or decrease in BP of 20 mmHg of patient's baseline BP within 5 minutes of endotracheal intubation will be considered significant in our study.

CONTACTS AND LOCATIONS:
Overall Officials: Warisha ismail Dr Warisha ismail, Principal Investigator — Liaquat National Hospital and Medical College
Locations (1):
- Liaquat National Hospital and Medical College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
*Informed consent*: Participants may not have provided informed consent for their data to be shared, which could raise ethical concerns.
  Patient confidentiality*: Sharing IPD could compromise patient confidentiality and anonymity, potentially harming participants or their families.
  IPD may require additional validation and quality control checks before sharing, which can be time-consuming and resource-intensive.

REFERENCES:
- See also: Kore SS, Teresa Jose VS, Shah KS. Therapeutic Efficacy of dexmedetomidine on the pressor response due to endotracheal intubation and on the induction dose of propofol for surgeries under general anesthesia — http://www.mjdrdypv.org